CLINICAL TRIAL: NCT01712841
Title: A Prospective Study Examining Patients With Non-exudative Age-related Macular Degeneration (NEAMD) of Different Severity
Brief Title: Non-exudative Age-related Macular Degeneration
Acronym: NEAMD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Thomas S. Hwang, MD, Associate Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: OHSU IRB #00008749
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Non-exudative Age-related Macular Degeneration
Keywords: Dry AMD; Age-related macular degeneration; Optical coherenece tomography; Imaging; Blood flow
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Severe NEAMD: Presence of definite central or noncentral geographic atrophy within 3000 microns of the foveal center
- Moderate/Intermediate NEAMD: Presence of large drusen (>125µ) and pigmentary changes without geographic atrophy
- Mild/Early NEAMD: Presence of small or medium drusen without geographic atrophy

SUMMARY:
Age-related macular degeneration (AMD) is the most prevalent cause of vision loss in developed countries and is often discussed in terms of the "dry" and the "wet" forms. The "wet" form of AMD is the more advanced form of the disease and is responsible for 80% of the legal blindness in AMD. Treatment options include a promising class of biologics called anti-vascular endothelial growth factors, as well as photodynamic therapy and laser surgery. These therapies can slow further vision loss, but cannot achieve recovery of lost vision. The "wet" form of AMD is always preceded by the "dry" form. Therefore, it is reasonable to expect that the early detection and treatment of the "dry" form may help reduce vision loss or progression to the more damaging "wet" form. Unfortunately, symptoms appear only in advanced stages of the "dry" form. As light sensitive cells in the macula breakdown in a process called geographic atrophy, the patient may notice blurred central vision.

OCT is an imaging technology that can perform non-contact cross-sectional imaging of retinal and choroidal tissue structure in real time. It is analogous to ultrasound B-mode imaging, except that OCT measures the intensity of reflected light rather than acoustical waves.

This study aims is to use OCT technology to compare how the retinal anatomy and blood flow differ within three severity groupings of non-exudative age-related macular degeneration (NEAMD).

ELIGIBILITY:
Inclusion Criteria:

* Presence of mild, moderate or severe NEAMD.
* Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs.
* Vision better than 20/200

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* A concurrent ocular pathology that may contribute to vision loss (e.g., CNV, glaucoma, visually significant cataract, optic neuropathy, diabetic retinopathy, history of retinal surgery) or interfere with acquisition of high-quality images
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* An ocular condition is present that, in the opinion of the investigator, might affect or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* Unable to ambulate and take tram from clinic to where OCT is located

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 60 and 85 years of age presenting to the Retina Service within the Department of Ophthalmology at the Casey Eye Institute of Oregon Health & Science University with signs and symptoms of non-exudative AMD.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with severe NEAMD who have changes in retinal anatomy/blood flow compared with patients with mild and moderate NEAMD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Hwang, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States